CLINICAL TRIAL: NCT03902964
Title: Needs Assessment After Cancer in Patients Treated for Breast Cancer
Acronym: EACE
Status: Completed | Type: Observational
Sponsor: Institut Jean-Godinot (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02191-54
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Breast Neoplasm Female; Quality of Life; Fear Cancer
MeSH Terms: conditions — Pathophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women treated for breast cancer in 2017 (cohort A): all patients who completed breast cancer treatment between January 1 and May 31, 2017. Withdrawal of men, metastatic patients from the outset, patients with a history of breast cancer or any other location, selection of 20 patients with breast cancer in situ at random
- women treated for breast cancer in 2015 (cohorte B): all patients who completed breast cancer treatment between January 1 and 31 May 2015. Withdrawal of men, metastatic patients from the outset, patients with a history of breast cancer or any other location, selection of 20 patients with breast cancer in situ at random

SUMMARY:
observational monocentric study

DETAILED DESCRIPTION:
observational monocentric study

Primary objective :

Describe post-cancer supportive care needs, assessed by questionnaire in patients treated for breast cancer after completion of treatment and 2 years later.

Secondary objective :

* Correlation between needs after cancer and the fear of recidivism assessed by the scale of the inventory of fear.
* Compare the need for supportive care between the end of treatment and 2 years after.
* Assess needs after cancer according to the stage of the disease
* Evaluate the needs after cancer according to the treatments received: surgery-radiotherapy versus surgery-chemotherapy-radiotherapy.
* Assess needs after cancer according to age and socio-professional category.

Schedule :

The selected patients then received a letter including an information and non-objection note, the post-cancer needs questionnaire, the Fear Inventory severity subscale questionnaire, and the QLQ-C30 questionnaire. A delay of 1 month was chosen to return the questionnaire with a phone call after 15 days for an analysis of responses in February 2019.

ELIGIBILITY:
Inclusion Criteria:

Women who have been treated for breast cancer and whose treatment ended in 2017 (cohort A) and in 2015 (cohort B), aged between 18 and 80 years, and who declared their non-opposition free and enlightened.

Exclusion Criteria:

Patients who have been treated for recurrence or 2nd cancer, metastases from the outset, male, refusal to participate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who completed breast cancer treatment between January 1 and May 31, 2017, and between January 1 and 31 May 2015. Withdrawal of men, metastatic patients from the outset, patients with a history of breast cancer or any other location, selection of 20 patients with breast cancer in situ at random in each of the 2 cohorts.
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Post-cancer needs analysis | 2 years
  Post-cancer needs analysis based on the "post-cancer needs assessment" questionnaire for patients in both cohorts

CONTACTS AND LOCATIONS:
Overall Officials: stephanie SERVAGI VERNAT, MD, Principal Investigator — Institut Jean-Godinot
Locations (1):
- Institut Jean Godinot, Reims, France

IPD SHARING:
Plan to Share IPD: No